CLINICAL TRIAL: NCT03909594
Title: Ultrasound Guided Fascia Iliaca Nerve Block With Bupivacaine and Adjuvant Ketamine vs. Bupivacaine Alone in Patients With Hip or Femur Fracture: a Double Blind Randomized Clinical Trial (BupiKet)
Brief Title: Bubiket Study: Ultrasound Guided Fascia Iliaca Nerve Block With Bupivacaine and Adjuvant Ketamine vs. Bupivacaine Alone
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The COVID Pandemic delayed start of study and currently the investigators are not interested in conducting the study.
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager; Co-Investigator, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-08-05
Record Dates: First submitted 2019-04-04; First posted 2019-04-10 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Pain, Musculoskeletal
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Bupivacaine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a randomized double blind study - - All the pharmacist and research manager
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nerve Block with Bupivacaine an (Experimental): Patients will receive an ultrasound guided regional nerve block with Bupivacaine (0.5% or 5 mg/ml) 2.5 mg/kg (max dose 175 kg) + Ketamine (50 mg/ml) 2 mg/kg. Each patient will be given a volume of 40 mL - this will be a mixture of Bupivacaine, Ketamine and 0.9% NS to make up the full 40 ml.
  Interventions: Drug: Bupivacaine; Drug: Ketamine
- Nerve Block with Bupivacaine al (Active Comparator): Patients will receive an ultrasound guided regional nerve block with Bupivacaine 0.5% only. Each patient will be given a volume of 40 ml - this will be a mixture of Bupivacaine and 0.9% NS to make up the full volume of 40 mL
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine
Drug: Ketamine — Ketamine
  Arms: Nerve Block with Bupivacaine an

SUMMARY:
The project is meant to evaluate the effect of a combination of medications (Bupivacaine + Ketamine) used in an ultra-sound guided nerve block for patients presenting to the Emergency Department (ED) with hip and/or femur fractures. The goal is to see whether the combination of these two medications will result in greater and longer-lasting pain relief, longer-lasting motor and sensory block and overall less need for opioid rescue analgesia.

DETAILED DESCRIPTION:
STUDY DESIGN

Subjects: Patients aged 18 years and older with isolated hip or femur fracture confirmed on x-ray.

DESIGN:

A randomized double-blind prospective superiority trail.

* Each patient will receive Morphine for analgesia prior to regional nerve block.

  * Patients < 65 years will receive Morphine 0.1 mg/kg every four hours as needed for 2 doses
  * Patients > 65 years will receive Morphine 0.05 mg/kg every four hours as needed for 2 doses
* Treatment group: will receive an ultrasound guided regional nerve block with Bupivacaine (0.5% or 5 mg/ml) 2.5 mg/kg (max dose 175 kg) + Ketamine (50 mg/ml) 2 mg/kg. Each patient will be given a volume of 40 mL - this will be a mixture of Bupivacaine, Ketamine and 0.9% NS to make up the full 40 ml.
* Control group: will receive an ultrasound guided regional nerve block with Bupivacaine 0.5% only. Each patient will be given a volume of 40 ml - this will be a mixture of Bupivacaine and 0.9% NS to make up the full volume of 40 mL
* The patients will be followed with respect to accrual time, follow up time, and total time of the block as well as a need for rescue analgesia as follows: every 15 minutes for the first hour; every 30 minutes for the next hour; every 1 hour for next 4 hours; every 4 hours for next 18 hours with end point of 24 hours or up until they are taken to surgery, whichever comes first.
* Evaluation of the sensory blocks: will be performed every 5 minutes after administration of the local anesthetic. The sensory block will be quantified as: 0 = Anesthesia (no sensation), 1 = Analgesia (decreased [dull] sensation), and 2 = no block (normal sensation), by using the pinprick test and comparing with the contralateral limb. The time elapsed from the injection to the onset of analgesia in the central sensory region of femoral nerve block will be taken as time of onset of the sensory block.
* Rescue Analgesia: If pain is not relieved and the participant requires rescue analgesia a weight-based dose of Morphine will be given at 0.1 mg/kg.

In addition, an antidote (lipid emulsion) that will be given to patients who need it when they develop severe side effects.

DATA COLLECTION:

Patient demographic, clinical and injury information, pain score, onset of motor and sensory block, rescue analgesia and side effects/adverse events will be collected by using a data collection form by trained research assistant and associates.

DATA ANALYSIS:

Statistical Analyses will include frequency distributions, t-test and chi-square for comparison between and within the groups and Cox Linear Regression Analysis. P<.05 will denote statistical significance. Statistical analyses will be conducted via SPSS version 24. Antonios Likourezos or equivalent will perform the statistical analyses.

EXPECTED OUTCOMES:

PRIMARY OUTCOME: time to first rescue analgesia post-regional nerve blockade in each group

SECONDARY OUTCOMES:

• Change in pain score as measured by Visual Analog Scale: Patient to be approached at the following intervals: every 15 minutes for the first hour; every 30 minutes for the next hour; every 1 hour for next 4 hours; every 4 hours for next 18 hours with end point of 24 hours or up until they are taken to surgery, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Presenting with isolated hip or femur fracture confirmed on x-ray.

Exclusion Criteria:

* Polytrauma
* Unstable vitals signs
* Allergy to Bupivacaine or Ketamine
* Inability to give consent
* Altered mental status
* Greater than 100kg
* Known end stage renal disease or hepatic dysfunction
* Received > 2 doses of Morphine in ER prior to regional nerve block
* Patients with failed nerve block (30 minute onset)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
time to first rescue analgesia post-regional nerve blockade | 0-24 hours
  The difference in time from administration of pain medication to rescue analgesia

SECONDARY OUTCOMES:
Pain score at 30 minutes | 30 minutes
  The pain score at 30 minutes at an 11 point Likert Numeric Rating Scale (0 = no pain; 5=moderate pain, and 10 = very severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Motov, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT03909594/Prot_SAP_000.pdf